CLINICAL TRIAL: NCT00171210
Title: An Extension Study of Iron Chelation Therapy With Deferasirox (ICL670)in β-thalassemia Patients With Transfusional Iron Overload
Brief Title: An Extension Study of Iron Chelation Therapy With Deferasirox (ICL670) in β-thalassemia Patients With Transfusional Iron Overload
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0107E1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Transfusional Iron Overload in β-thalassemia
Keywords: β-thalassemia; iron overload; deferasirox
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): All participants received Deferasirox (ICL670) orally once a day. Dosage based on body weight.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Tablets taken orally once a day.

SUMMARY:
A 1-year randomized Phase III core trial (NCT00061750) using deferoxamine as the comparator was conducted to investigate the efficacy of deferasirox in regularly transfused patients with β-thalassemia 2 years of age and older. Patients who successfully completed this main trial may continue in this extension trial to receive chelation therapy with deferasirox for an additional 4 years.

The objective of this study is to assess the efficacy and long-term safety of deferasirox in regularly transfused patients with β-thalassemia 2 years of age and older.

ELIGIBILITY:
Inclusion criteria

* Patients who completed the 12-month core study (NCT00061750)
* Female patients after menarche and who were sexually active, if they used double-barrier contraception, oral contraceptive plus barrier contraceptive, or had undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation
* Written informed consent obtained from the patient and/or legal guardian on the patient's behalf in accordance with the national legislation

Exclusion criteria

* Pregnant or breast feeding patients
* Patients with a history of non-compliance to medical regimens or those considered to be potentially unreliable

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Stanford Hospital, Division of Oncology, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital Boston, Dept of Hematology, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mons
- Brazil (2):
  - Novartis Investigative Site, Campinas
  - Novartis Investigative Site, São Paulo
- Canada (2):
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Toronto
- France (4):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Italy (14):
  - Novartis Investigative Site, Brindisi
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Ferrara
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Naples
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Sassari
  - Novartis Investigative Site, Syracuse
  - Novartis Investigative Site, Turin
- Novartis Investigative Site, Tunis, Tunisia
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Isparta
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Cappellini MD, Bejaoui M, Agaoglu L, Canatan D, Capra M, Cohen A, Drelichman G, Economou M, Fattoum S, Kattamis A, Kilinc Y, Perrotta S, Piga A, Porter JB, Griffel L, Dong V, Clark J, Aydinok Y. Iron chelation with deferasirox in adult and pediatric patients with thalassemia major: efficacy and safety during 5 years' follow-up. Blood. 2011 Jul 28;118(4):884-93. doi: 10.1182/blood-2010-11-316646. Epub 2011 May 31. PMID 21628399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is an extension of core study (NCT0061750). 555 participants were treated with Deferasirox (ICL670) in the core and/or extension study. In the core study, 296 participants were treated with ICL670 and 259 participants were treated with Deferoxamine(DFO).
Groups:
- Crossover: Participants treated with Deferoxamine (DFO) during the core study and crossed over to receive Deferasirox (ICL670) orally once a day during the extension study. Dosage based on body weight.
- ICL670: Participants treated with Deferasirox (ICL670) orally once a day during the core study and continued this treatment in the extension study. Dosage based on body weight.
Period: Overall Study
Arm/Group | Crossover | ICL670
Started | 259 | 296
STARTED EXTENSION STUDY | 259 | 247
Completed | 190 | 181
Not Completed | 69 | 115
Not completed — Adverse Event | 16 | 27
Not completed — Abnormal laboratory value(s) | 6 | 3
Not completed — Abnormal test procedure result(s) | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 11 | 15
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 32 | 30
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 1 | 1
Not completed — Death | 2 | 3
Not completed — Stopped at end of core | 0 | 32
Not completed — Stopped at end of extension 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover | ICL670 | Total
Number analyzed (Participants) | 259 | 296 | 555
Age Continuous [Mean (Standard Deviation); unit: years] | 18.3 (9.82) | 17.1 (9.46) | 17.7 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 156 | 281
  Male | 134 | 140 | 274
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 2 | 3
  White | 225 | 263 | 488
  Oriental | 10 | 9 | 19
  Other | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety and Tolerability Profile of ICL670 Based on the Number of Participants Who Experienced Any Adverse Event
Description: Adverse events results are based on preferred terms with at least 7% of participants in any group.
Time Frame: up to 5 years
Population: All patients enrolled into core study and who consented to participate in extension contributed to the pool of data on long term safety follow-up. Analyses included all patients who received at least 1 dose of ICL670 in the core/extension study, that is, analyses also included ICL670 patients from the core group who did not continue into extension.
Measure: Number; unit: Participants
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 259 | 296
Participants
  Pyrexia | 109 | 113
  Cough | 85 | 110
  Headache | 81 | 84
  Diarrhoea | 73 | 69
  Vomiting | 61 | 75
  Influenza | 65 | 70
  Abdominal pain | 59 | 75
  Nasopharyngitis | 56 | 73
  Nausea | 52 | 63
  Oropharyngeal pain | 50 | 62
  Pharyngitis | 57 | 55
  Back Pain | 49 | 59
  Abdominal pain upper | 52 | 52
  Rhinitis | 45 | 52
  Bronchitis | 41 | 45
  Arthralgia | 39 | 45
  Upper respiratory tract infection | 32 | 52
  Transfusion reaction | 36 | 34
  Blood creatinine increased | 22 | 47
  Gastroenteritis | 31 | 37
  Asthenia | 31 | 31
  Rash | 24 | 34
  Tonsillitis | 22 | 30
  Fatigue | 22 | 29
  Pain in extremity | 21 | 30
  Acute tonsillitis | 21 | 29
  Dyspepsia | 17 | 21
  Urinary tract infection | 14 | 23
  Urticaria | 14 | 23
  Toothache | 14 | 22
  Sinusitis | 13 | 22
  Cholelithiasis | 11 | 23

2. Secondary Outcome: Long-term Effect of ICL670 on Hepatic Iron Stores Measured by Means of Liver Iron Content (LIC) as Assessed by Liver Biopsy
Description: Mean absolute change of LIC from start of Deferasirox (ICL670) treatment to the end of study assessed by liver biopsy. Reported in milligrams of Iron per gram dry weight (mg Fe/g dw).
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: Population includes only those participants from the full analysis set (defined as all participants who received at least 1 dose of ICL670 in the core/extension study, that is, analyses also included ICL670 participants from the core group who did not continue into extension) and had LIC Biopsy data at Start of ICL670 treatment and End of Study.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 95 | 220
mg Fe/g dw | -2.4 (8.23) | -4.1 (10.31)

3. Secondary Outcome: Long-term Effect of ICL670 on Hepatic Iron Stores Measured by Means of Liver Iron Content (LIC) as Assessed by SQUID
Description: Mean absolute change in LIC from start of Deferasirox (ICL670) treatment to the end of the study assessed by Superconducting Quantum Interfering Device (SQUID) measurement used as a non-invasive alternative to Biopsy for pediatric participants. Reported in milligrams of Iron per gram dry weight (mg Fe/g dw).
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: Population includes only those participants from the full analysis set (defined as all participants who received at least 1 dose of ICL670 in the core/extension study, that is, analyses also included ICL670 participants from the core group who did not continue into extension) and had LIC SQUID data at Start of ICL670 treatment and End of Study.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 34 | 44
mg Fe/g dw | -0.5 (5.34) | -0.7 (4.03)

4. Secondary Outcome: Long-term Effect of Treatment With ICL670 on the Changes in Serum Ferritin Levels From Start of ICL670 Treatment to End of Study
Description: Mean Absolute Change in serum ferritin (ug/L) from start of treatment with Deferasirox (ICL670) to end of study taking into account the therapeutic goal which will either be to maintain iron balance or to induce negative iron balance. End of study taken as the mean of, at most, the last three available results after start of treatment with ICL670.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 259 | 296
μg/L | -122.1 (1406.77) | -527.8 (1852.12)

5. Secondary Outcome: Change in Surrogate Marker: Serum Transferrin From Start of Treatment With ICL670 to End of Study
Description: Measurement of the relative change in percent of potential surrogate marker: Serum Transferrin (g/L) from start of treatment with Deferasirox (ICL670) to end of study.
  (Serum Transferrin at the End of Study-Serum Transferrin at Start of ICL670)/Serum Transferrin at Start of ICL670*100.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 259 | 296
Percent change | 7.7 (16.3) [-4.6 to 0.1] | 7.0 (14.78) [-4.6 to 0.1]

6. Secondary Outcome: Change in Surrogate Marker: Serum Iron From Start of Treatment With ICL670 to End of Study
Description: Measurement of the relative change of potential surrogate markers: Serum Iron (µmol/L) from start of treatment with Deferasirox (ICL670) to end of study.
  (Serum Iron at the End of Study-Serum Iron at Start of ICL670)/Serum Iron at Start of ICL670*100.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 259 | 296
Percent change | 1.5 (29.99) | 10.3 (39.07)

7. Secondary Outcome: Change in Surrogate Marker: Transferrin Saturation From Start of Treatment With ICL670 to End of Study
Description: Measurement of the relative change of potential surrogate marker: Transferrin Saturation (Percent) from start of treatment with Deferasirox (ICL670) to end of study.
  (Transferrin Saturation at the End of Study-Tranferrin Saturation at Start of ICL670)/Transferrin Saturation at Start of ICL670*100.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 259 | 296
Percent change | -5.4 (27.06) | 3.4 (36.17)

8. Secondary Outcome: Absolute Change in Liver Iron Content From Start of ICL670 Treatment to End of Study Measured by Biopsy
Description: Measurement of median absolute change in liver iron content (LIC) from start of treatment with Deferasirox (ICL670) to end of study obtained through biopsy. Absolute change = End of study value - start of treatment value. LIC is expressed in mg of iron per gram of liver dry weight (mg Fe/g dw).
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 2
Measure: Median (Full Range); unit: mg Fe/g dw
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 95 | 220
mg Fe/g dw | -2.8 (8.23) [-24.0 to 18.4] | -3.2 (10.31) [-34.7 to 31.4]

9. Secondary Outcome: Relative Change in Liver Iron Content From Start of ICL670 Treatment to End of Study Measured by Biopsy
Description: Relative change in liver iron content (LIC) as measured by biopsy and calculated by: End of study value - Start of ICL670 treatment value (absolute change) / Start of ICL670 treatment value.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 2
Measure: Median (Full Range); unit: percent of start value
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 95 | 220
percent of start value | -25.4 [-97.6 to 314.6] | -26.0 [-100.0 to 581.5]

10. Secondary Outcome: Absolute Change in Liver Iron Content From Start of ICL670 Treatment to End of Study Measured by SQUID
Description: Measurement of the median absolute change in liver iron content (LIC) from start of treatment with Deferasirox (ICL670) to end of study obtained through Superconducting Quantum Interfering Device (SQUID). Absolute change = End of study value - start of treatment value. LIC is expressed in mg of iron per gram of liver dry weight (mg Fe/g dw).
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 3
Measure: Median (Full Range); unit: mg Fe/g dw
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 34 | 44
mg Fe/g dw | -1.1 [-14.1 to 18.1] | -1.6 [-8.7 to 12.0]

11. Secondary Outcome: Relative Change in Liver Iron Content From Start of ICL670 Treatment to End of Study as Measured by SQUID
Description: Relative change in liver iron content (LIC) measured by Superconducting Quantum Interfering Device (SQUID), calculated by: End of study value - Start of ICL670 treatment value (absolute change) / Start of ICL670 treatment value.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 3
Measure: Median (Full Range); unit: percent of start value
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 34 | 44
percent of start value | -20.8 [-84.4 to 517.1] | -33.0 [-87.0 to 218.2]

12. Secondary Outcome: Change of Total Body Iron Excretion Rate (TBIE) From Start of ICL670 Treatment to the End of Study
Description: Median change in TBIE (mg/kg/day) from start of treatment with Deferasirox (ICL670) to end of study.
Time Frame: Start of ICL670 treatment, End of Study or study discontinuation (up to 5 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | Crossover | ICL670
Number analyzed (Participants) | 129 | 266
mg/kg/day | 0.37 [0.07 to 0.78] | 0.38 [-0.14 to 1.00]

ADVERSE EVENTS:
Groups:
- ICL670: Participants treated with Deferasirox (ICL670) orally once a day during the core study continued this treatment in the extension study. Dosage based on body weight.
Arm/Group | ICL670 | Crossover
Serious Adverse Events (participants affected / at risk) | 102/296 | 61/259
Other Adverse Events (participants affected / at risk) | 266/296 | 236/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=296) | Crossover (N=259)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 5 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Accessory spleen (Congenital, familial and genetic disorders) | 0 | 1
Thalassaemia beta (Congenital, familial and genetic disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Lenticular opacities (Eye disorders) | 1 | 1
Papilloedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 2
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 3 | 0
Chest pain (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 6
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 7 | 6
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 3 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
HIV infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Yersinia infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Cardiovascular function test abnormal (Investigations) | 0 | 1
Cells in urine (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Serum ferritin increased (Investigations) | 0 | 1
Streptococcal identification test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Clumsiness (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 0
Glomerulonephropathy (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Splenectomy (Surgical and medical procedures) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=296) | Crossover (N=259)
Palpitations (Cardiac disorders) | 17 | 11
Ear pain (Ear and labyrinth disorders) | 16 | 14
Abdominal pain (Gastrointestinal disorders) | 74 | 57
Abdominal pain upper (Gastrointestinal disorders) | 51 | 52
Constipation (Gastrointestinal disorders) | 17 | 13
Diarrhoea (Gastrointestinal disorders) | 68 | 73
Dyspepsia (Gastrointestinal disorders) | 21 | 17
Nausea (Gastrointestinal disorders) | 62 | 52
Toothache (Gastrointestinal disorders) | 22 | 14
Vomiting (Gastrointestinal disorders) | 72 | 61
Asthenia (General disorders) | 29 | 31
Fatigue (General disorders) | 29 | 22
Influenza like illness (General disorders) | 12 | 17
Oedema peripheral (General disorders) | 17 | 15
Pyrexia (General disorders) | 110 | 108
Cholelithiasis (Hepatobiliary disorders) | 18 | 5
Acute tonsillitis (Infections and infestations) | 28 | 21
Bronchitis (Infections and infestations) | 42 | 41
Ear infection (Infections and infestations) | 22 | 7
Gastroenteritis (Infections and infestations) | 37 | 29
Influenza (Infections and infestations) | 70 | 65
Nasopharyngitis (Infections and infestations) | 73 | 56
Pharyngitis (Infections and infestations) | 54 | 57
Rhinitis (Infections and infestations) | 52 | 45
Sinusitis (Infections and infestations) | 21 | 13
Tonsillitis (Infections and infestations) | 29 | 22
Tooth abscess (Infections and infestations) | 15 | 8
Upper respiratory tract infection (Infections and infestations) | 52 | 32
Urinary tract infection (Infections and infestations) | 23 | 14
Transfusion reaction (Injury, poisoning and procedural complications) | 32 | 36
Blood creatinine increased (Investigations) | 46 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 59 | 49
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 17 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 20
Headache (Nervous system disorders) | 84 | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 110 | 85
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 62 | 50
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Rash (Skin and subcutaneous tissue disorders) | 33 | 24
Urticaria (Skin and subcutaneous tissue disorders) | 23 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.